CLINICAL TRIAL: NCT04106765
Title: Clinical, EEG and Radiological Initial and Evolutive Characterisation of LGI1-antibody Patients
Brief Title: LGI1-antibody Patients Follow-up
Acronym: evoLGI1
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: evoLGI1
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-09

CONDITIONS: Anti-LGI1 Encephalitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- : epileptic LGI1-antibody patients: Patients affected by LGI1 antibody encephalitis presenting epileptic seizures as a first symptom
  Evaluated items:
  * Number of seizures
  * Type of seizures
  * Presence of EEG abnormalities
  * Presence of IRM abnormalities
  * Time before cognitive disorders
- cognitive LGI1-antibody patients: Patients affected by LGI1 antibody encephalitis presenting cognitive disorders as a first symptom
  Evaluated items:
  * Presence of EEG abnormalities
  * Presence of IRM abnormalities
  * Time before epileptic seizures

SUMMARY:
Autoimmune encephalitis involve autoantibodies targeting central nervous system, and particularly the synapse or its structure like for LGI1 protein. Anti-LGI1 encephalitis is revealed by an inflammation of the limbic system, with mainly temporal lobe, faciobrachial dystonic or generalized seizures, and cognitive disorders.

This disease is rare and its clinical, EEG and radiological characterisation is not sufficiently established. The investigators will evaluate these three aspects for the anti-LGI1 cohort of patients of the National Reference Center of autoimmune encephalitis.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Diagnosis of anti-LGI1 encephalitis based on sera or CSF samples in the National Reference Center of autoimmune encephalitis from 2011/06 to 2019 july 1st.
* Clinical follow-up in France

Exclusion Criteria:

* Anti-LGI1 antibody associated with another encephalitis antibody
* Foreign follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study Population Description : Adult patients presenting an anti-LGI1 autoimmune encephalitis, followed in France and diagnosed by sera or CSF samples at the National Reference Center of autoimmune encephalitis.
Sampling Method: Non-Probability Sample
Enrollment: 192 (Estimated)
Dates: Start 2019-10-30 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Evolution of epileptic seizures | 12 MONTHS

CONTACTS AND LOCATIONS:
Overall Officials: Jerome HONNORAT, pHd, Principal Investigator — National Reference Center of autoimmune encephalitis
Locations (1):
- Centre de référence des syndromes neurologiques paranéoplasiques et encéphalites auto-immunes, Lyon, France

IPD SHARING:
Plan to Share IPD: No